CLINICAL TRIAL: NCT01122654
Title: Growth and Tolerance of Cow Milk-Based Infant Formulas
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Tim Cooper, M.D., Mead Johnson Nutrition
Other Study IDs: 3380-1
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control
- Experimental 1
- Experimental 2

SUMMARY:
This clinical trial will assess growth, tolerance and adverse events of cow milk-based infant formulas in healthy, term infants.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 12-16 days of age at randomization
* Term infant with birth weight of minimum of 2500 g
* Solely formula fed
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* History of underlying metabolic or chronic disease or immunocompromised
* Acute infection
* Feeding difficulties or formula intolerance

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy, term infants
Sampling Method: Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Body weight measured on calibrated infant scale at each study visit

SECONDARY OUTCOMES:
Twenty-four hour recall of infant formula intake at each study visit
Medically-confirmed adverse events collected throughout the study period
Twenty-four hour recall of stool characteristics (number and consistency) and tolerance at each study visit
Parental Product Assessment Questionnaire completed at Study Visit 2
  Assessment of physical properties of product and infant's reaction during consumption.
Body Length and Head Circumference measured at each study visit

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Pediatrics East - Alabama Clinical Therapeutics, Pinson, Alabama
  - Central Arkansas Pediatric Clinic, Benton, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Altamonte Pediatric Associates, Lake Mary, Florida
  - Children's Medical Association, Plantation, Florida
  - North Georgia Clinical Research Center/White's Pediatrics, Dalton, Georgia
  - Deaconess Clinic Gateway, Newburgh, Indiana
  - PTCU/Children & Youth Project, Louisville, Kentucky
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Southwestern Medical Clinic, PC, Niles, Michigan
  - Southwestern Medical Clinic P.C., Stevensville, Michigan
  - The Center for Human Nutrition, Omaha, Nebraska
  - Cary Pediatric Center, PA, Cary, North Carolina
  - Innovis Health South University, Fargo, North Dakota
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - Alpha Clinical Research, Clarksville, Tennessee
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Austin Diagnostic Clinic, Austin, Texas

REFERENCES:
- [Derived] Johnston WH, Ashley C, Yeiser M, Harris CL, Stolz SI, Wampler JL, Wittke A, Cooper TR. Growth and tolerance of formula with lactoferrin in infants through one year of age: double-blind, randomized, controlled trial. BMC Pediatr. 2015 Nov 7;15:173. doi: 10.1186/s12887-015-0488-3. PMID 26547414